CLINICAL TRIAL: NCT02511353
Title: Efficacy and Safety of High-dose Ivermectin for Reducing Malaria Transmission: A Dose Finding Study (IVERMAL)
Brief Title: Efficacy and Safety of High-dose Ivermectin for Reducing Malaria Transmission: A Dose Finding Study
Acronym: IVERMAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Kenya Medical Research Institute (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14.002; 2775 (Other: Kenya Medical Research Institute); 6720 (Other: Centers for Disease Control and Prevention)
Record Dates: First submitted 2015-07-15; First posted 2015-07-30 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Malaria
Keywords: malaria; plasmodium; dihydroartemisinin-piperaquine; ivermectin
MeSH Terms: conditions — Malaria | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): Standard 3-day course of dihydroartemisinin-piperaquine, plus once a day for 3 days: placebo 600 mcg/kg/day.
  Interventions: Drug: placebo; Drug: dihydroartemisinin-piperaquine
- ivermectin 300 mcg/kg (Experimental): Standard 3-day course of dihydroartemisinin-piperaquine, plus once a day for 3 days: ivermectin 300 mcg/kg/day and placebo 300 mcg/kg/day.
  Interventions: Drug: ivermectin; Drug: placebo; Drug: dihydroartemisinin-piperaquine
- ivermectin 600 mcg/kg (Experimental): Standard 3-day course of dihydroartemisinin-piperaquine, plus once a day for 3 days: ivermectin 600 mcg/kg/day.
  Interventions: Drug: ivermectin; Drug: dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: ivermectin
  Arms: ivermectin 300 mcg/kg; ivermectin 600 mcg/kg
Drug: placebo — Placebo for ivermectin.
  Arms: ivermectin 300 mcg/kg; placebo
Drug: dihydroartemisinin-piperaquine

SUMMARY:
In western Kenya the prevalence of malaria in <5 year olds has fallen from 70% in 1997 to 40% in 2008, where it has now stagnated. Innovative approaches are needed to continue towards elimination. Ivermectin is a broad spectrum antiparasitic endectocide widely used for the control of onchocerciasis and lymphatic filariasis at a dose of 150-200 mcg/kg. Ivermectin at this dose has a potent, but short-lived effect for 6-11 days on mosquito survival, egg-laying, and parasite sporogony. Higher doses are needed to prolong its mosquitocidal effects. Previous studies have shown ivermectin is very well tolerated and safe even up to 2,000 mcg/kg. This dose finding study will evaluate the transmission blocking effect of high-dose ivermectin to define the optimal dose for future use of ivermectin in combination with artemisinin-based combination therapy (ACT) for mass drug administration (MDA). It explores a research question of global relevance. A prolonged transmission blocking effect of ivermectin could have substantial consequences for malaria control in the next decades. The results are expected to inform national malaria control programs in malaria endemic countries, to inform WHO guidelines, and to contribute to the regulatory process.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic, uncomplicated Plasmodium falciparum infection
* Positive malaria microscopy or malaria RDT (pLDH)
* Age: 18-50 years
* Provide written informed consent
* Agree to be able to travel to clinic on days: 1, 2, 7, 10, 14, 21, and 28

Exclusion Criteria:

* Signs or symptoms of severe malaria
* Unable to provide written informed consent
* For women: pregnancy or lactation
* Hypersensitivity to ivermectin or DP
* QTc >460 ms on ECG
* Body Mass Index (BMI) below 16 or above 32 kg/m2
* Haemoglobin concentration below 9 g/dL
* Taken ivermectin in the last month
* Taken dihydroartemisinin-piperaquine in the last 12 weeks
* Loa loa as assessed by travel history to Angola, Cameroon, Chad, Central African Republic, Congo, DR Congo, Equatorial Guinea, Ethiopia, Gabon, Nigeria and Sudan
* History and/or symptoms indicating chronic illness
* Current use of tuberculosis or anti-retroviral medication
* Previously enrolled in the same study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Mosquito survival | Survival of mosquitoes at 14 days after feeding on blood taking from study participants who started the 3-day ivermectin and DP regimen 7 days earlier.

SECONDARY OUTCOMES:
Mosquito survival | Survival of mosquitoes at each day up to day 21 or 28 after each feeding experiments performed at 0, 2 day+4h, 10, 14, 21, 28 days after start of treatment.
Number of patients with malaria clinical and parasitological treatment response | Up to day 28.
Area under the plasma concentration versus time curve (AUC) of ivermectin | Up to day 28.
Area under the plasma concentration versus time curve (AUC) of piperaquine | Up to day 28.
  Dihydroartemisinin-piperaquine is a combination drug. As dihydroartemisinin has a very short elimination time, only the AUC for the longer acting piperaquine component will be determined.
Peak plasma Concentration (Cmax) of ivermectin | Up to day 28.
Peak plasma Concentration (Cmax) of piperaquine | Up to day 28.
  Dihydroartemisinin-piperaquine is a combination drug. As dihydroartemisinin has a very short elimination time, only the Cmax for the longer acting piperaquine component will be determined.
Tolerability as assessed by adverse events reported in a general toxicity questionnaire | Up to day 28.
CNS adverse events | Up to day 28.
Serious adverse events | Up to day 28.
Haemoglobin concentrations | Up to day 28.
QTc interval | At 52 hours.
Mydriasis quantitated by pupillometry | Up to day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Menno R. Smit, MD, MPH, Principal Investigator — Liverpool School of Tropical Medicine; Feiko ter Kuile, Prof., Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- Jaramogi Oginga Odinga Teaching and Referral Hospital, Kisumu, Kenya

REFERENCES:
- [Background] Smit MR, Ochomo E, Aljayyoussi G, Kwambai T, Abong'o B, Bayoh N, Gimnig J, Samuels A, Desai M, Phillips-Howard PA, Kariuki S, Wang D, Ward S, Ter Kuile FO. Efficacy and Safety of High-Dose Ivermectin for Reducing Malaria Transmission (IVERMAL): Protocol for a Double-Blind, Randomized, Placebo-Controlled, Dose-Finding Trial in Western Kenya. JMIR Res Protoc. 2016 Nov 17;5(4):e213. doi: 10.2196/resprot.6617. PMID 27856406
- [Result] Smit MR, Ochomo EO, Aljayyoussi G, Kwambai TK, Abong'o BO, Chen T, Bousema T, Slater HC, Waterhouse D, Bayoh NM, Gimnig JE, Samuels AM, Desai MR, Phillips-Howard PA, Kariuki SK, Wang D, Ward SA, Ter Kuile FO. Safety and mosquitocidal efficacy of high-dose ivermectin when co-administered with dihydroartemisinin-piperaquine in Kenyan adults with uncomplicated malaria (IVERMAL): a randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2018 Jun;18(6):615-626. doi: 10.1016/S1473-3099(18)30163-4. Epub 2018 Mar 27. PMID 29602751
- [Result] Smit MR, Ochomo EO, Waterhouse D, Kwambai TK, Abong'o BO, Bousema T, Bayoh NM, Gimnig JE, Samuels AM, Desai MR, Phillips-Howard PA, Kariuki SK, Wang D, Ter Kuile FO, Ward SA, Aljayyoussi G. Pharmacokinetics-Pharmacodynamics of High-Dose Ivermectin with Dihydroartemisinin-Piperaquine on Mosquitocidal Activity and QT-Prolongation (IVERMAL). Clin Pharmacol Ther. 2019 Feb;105(2):388-401. doi: 10.1002/cpt.1219. Epub 2018 Oct 9. PMID 30125353
- [Derived] Smit MR, Ochomo EO, Aljayyoussi G, Kwambai TK, Abong'o BO, Bousema T, Waterhouse D, Bayoh NM, Gimnig JE, Samuels AM, Desai MR, Phillips-Howard PA, Kariuki SK, Wang D, Ward SA, Ter Kuile FO. Human Direct Skin Feeding Versus Membrane Feeding to Assess the Mosquitocidal Efficacy of High-Dose Ivermectin (IVERMAL Trial). Clin Infect Dis. 2019 Sep 13;69(7):1112-1119. doi: 10.1093/cid/ciy1063. PMID 30590537